CLINICAL TRIAL: NCT02090673
Title: Post-Marketing Surveillance Study: 12 To 24 Weeks Study On The Treatment Emergent Adverse Events In Patients With Type 2 Diabetes Taking Exenatide In Korea
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MB001-078
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group1:Type 2 diabetic patients treated with Exenatide therapy: Korean patients who are at least 18 years old, diagnosed with type 2 diabetes, and are treated with Exenatide in an ambulatory care setting according to the approved label
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide

SUMMARY:
The objective of this regulatory Post-Marketing Surveillance in Korea is to reconfirm the clinical usefulness of Exenatide through collecting, reviewing, identifying and verifying the safety and effectiveness information about Exenatide in general practice.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female at least 18 years of age
* Patients who are to initiate Exenatide treatment for type 2 diabetes at baseline, following their treating physicians' advice
* Patients, who in the opinion of the treating physicians, comply with all the recommendations stated in the relevant product information

Exclusion Criteria:

* Are simultaneously participating in a different study that includes a treatment intervention and/or an investigational drug
* Are pregnant or have intentions of becoming pregnant within the duration of the study
* Contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, hospital and teaching hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1711 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The proportion of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) in patients who are treated with Exenatide for type 2 diabetes mellitus | At 12 weeks ± 4 weeks or 24 weeks ± 4 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint in Hemoglobin A1c (HbA1c) | Baseline (Day 1) and 12 or 24 weeks ± 4 weeks
Change from baseline to endpoint in Body weight | Baseline (Day 1) and 12 or 24 weeks ± 4 weeks
Change from baseline to endpoint in Fasting plasma glucose | Baseline (Day 1) and 12 or 24 weeks ± 4 weeks
Change from baseline to endpoint in subjective measures include improvement of main indication | Baseline (Day 1) and 12 or 24 weeks ± 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- [Derived] Hwang YC, Kim A, Jo E, Yang Y, Cho JH, Lee BW. Effectiveness and safety of exenatide in Korean patients with type 2 diabetes inadequately controlled with oral hypoglycemic agents: an observational study in a real clinical practice. BMC Endocr Disord. 2017 Oct 25;17(1):68. doi: 10.1186/s12902-017-0220-4. PMID 29065865
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CSR_Synopsis_MB001-078.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3673&filename=CSR_Synopsis_MB001-078.pdf